CLINICAL TRIAL: NCT02593552
Title: Video Intervention to Enhance the Safety Of Cognitively Impaired Older Drivers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Brian Ott, Brian R. Ott, MD, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 263758-14
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Impaired Driving

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Video camera (Experimental): DriveCam video event recorder with counseling feedback
  Interventions: Device: DriveCam

INTERVENTIONS:
Device: DriveCam — Video event monitoring device

SUMMARY:
This pilot study was done to assess the feasibility and possible efficacy of a video feedback intervention to improve the safety of cognitively impaired older drivers.

DETAILED DESCRIPTION:
The goals of this pilot study were to demonstrate that 1) g-force technology can effectively detect unsafe driving events by older adults, and 2) cognitively impaired older adults can improve their driving safety with an in-car video feedback intervention. Unsafe driving events were triggered by g-forces leading to capture of a video record that was then transmitted wirelessly to a remote office where the events were analyzed and scored. During the baseline phase (3 months), there was no feedback. During the intervention phase (4-6 months), participants received a weekly progress report in the mail along with DVD of recorded unsafe driving events with recommendations. The research team then contacted the participant and informant weekly to provide additional coaching, and verify that participants reviewed the information and videos. During the post-intervention monitoring phase (7-9 months), there was no further feedback. The primary quantitative outcomes were total number of unsafe driving events/1,000 miles and total safety driving score/1,000 miles. Secondary qualitative outcomes included the types and severity of unsafe driving events that were recorded.

ELIGIBILITY:
Inclusion Criteria:

* age 60-90
* English speaking
* currently driving adults with a valid driving license and at least 10 years of driving experience
* neurological examinations judged to be normal for age or consistent with AD
* questionable to mild dementia (CDR 0.5 to 1)
* MMSE < 28
* have an adult family member or other caregiver, age >21 to participate in counseling feedback

Exclusion Criteria:

* ophthalmologic, physical, or neurologic disorders other than dementia that impair their driving abilities
* visual acuity worse than 20/40 in best eye using distance vision measured by wall chart
* homonymous hemianopia or bitemporal hemianopia on confrontation testing
* musculoskeletal disorders causing major physical handicaps such as frozen joints, inadequately healed fractures, and amputations
* history of alcohol or substance abuse by DSM V diagnostic criteria within the past year
* sedating medications that impair level of consciousness or attention
* language impairment that would interfere with the ability to participate in the educational intervention
* previous road test evaluation or opinion of caregiver or health professional that subject is unsafe to drive.

Ages: 68 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of unsafe driving events | 9 months
  Scale

SECONDARY OUTCOMES:
Severity score of unsafe driving events | 9 months
  Scale

REFERENCES:
- [Derived] Ott BR, Davis JD, Bixby K. Video Feedback Intervention to Enhance the Safety of Older Drivers With Cognitive Impairment. Am J Occup Ther. 2017 Mar/Apr;71(2):7102260020p1-7102260020p7. doi: 10.5014/ajot.2017.020404. PMID 28218593